CLINICAL TRIAL: NCT03819972
Title: The Dose Response of Milk Minerals High in Calcium With Protein on Plasma Glucagon-Like Peptide-1 Concentrations
Brief Title: The Dose Response of Calcium Co-ingested With Protein on GLP-1 Concentrations
Acronym: PROCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Collaborators: Arla Foods (Industry)
Responsible Party: Principal Investigator, Jonathan Watkins, PhD Student, University of Bath
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PROCAL-JW
Record Dates: First submitted 2019-01-21; First posted 2019-01-29 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: GLP-1 Concentration

STUDY DESIGN:
Intervention Model Description: There are 4 conditions where participants will ingest differing amounts of calcium in a randomised order
Who Masked: Participant, Investigator
Masking Description: Participant will not be told which drink they will ingest until the end of the study.
  Individuals not collaborating on the study will randomise the drink order and make up the drinks so the investigator is blinded to which drink the particpant will ingest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): Participants will ingest a drink containing 25 g whey protein hydrolysate (227 mg of total calcium ingested)
  Interventions: Dietary Supplement: Dose response of Capolac®
- Dose 1 (Active Comparator): Participants will ingest a drink containing 25 g whey protein hydrolysate and 3179 mg Capolac (984 mg of total calcium ingested)
  Interventions: Dietary Supplement: Dose response of Capolac®
- Dose 2 (Active Comparator): Participants will ingest a drink containing 25 g whey protein hydrolysate and 6363 mg Capolac (1742 mg of total calcium ingested)
  Interventions: Dietary Supplement: Dose response of Capolac®
- Dose 3 (Active Comparator): Participants will ingest a drink containing 25 g whey protein hydrolysate and 9547 mg Capolac (2500 mg of total calcium ingested)
  Interventions: Dietary Supplement: Dose response of Capolac®

INTERVENTIONS:
Dietary Supplement: Dose response of Capolac® — Capolac® (milk minerals high in calcium) dose is manipulated

SUMMARY:
Hormones that are produced by our stomach and intestines play a role in regulating our appetite and health. One of the most important hormones is called GLP-1. The food we eat influences the release of this hormone and evidence suggests that protein and calcium are key nutrients that stimulate the secretion of GLP-1. We want to know if there is a dose related response by increasing the amount of calcium ingested with a constant amount of protein on the release of this hormone. We hypothesise that with increasing calcium dose we will see an increase in GLP-1 concentrations in a curvilinear pattern. This may have benefits for prescribing an optimal dose of calcium for weight maintenance and health.

DETAILED DESCRIPTION:
Recent work at the University of Bath has shown that when ingested with 50 g whey protein hydrolysate, Capolac® (milk minerals high in calcium) potently stimulates availability of the important hormone glucagon-like peptide-1 (GLP-1). However, it is currently unknown as to whether there is a dose dependent response to calcium co-ingestion with protein. Therefore we aim to perform a study on the effect of co-ingesting different doses of Capolac® with 25 g whey protein hydrolysate on GLP-1 availability. This project will help identify the calcium dose required with a moderate amount of protein to optimise GLP-1 availability and also provide insight into whether this may affect food intake and appetite.

Twenty metabolically healthy men and women, age 18-65 years, BMI between 25 and 34.9 kg/m2 will be recruited to participate in a randomised crossover study. Each participant will undergo 4 trials. Each trial will last ~4 hours and will be separated by a minimum of 48h:

1. CONTROL - 25 g whey protein hydrolysate (227 mg of total calcium ingested)
2. DOSE 1 - 25 g whey protein hydrolysate + 3179 mg Capolac (984 mg of total calcium ingested)
3. DOSE 2 - 25 g whey protein hydrolysate + 6363 mg Capolac (1742 mg of total calcium ingested)
4. DOSE 3 - 25 g whey protein hydrolysate + 9547 mg Capolac (2500 mg of total calcium ingested) Each of these drinks will also contain 500 mL of water and low calorie sweetener (80 mg sucralose).

Participants will be asked to arrive to the laboratory between 08:00 and 9:00 am after not eating for between 10-14 hours i.e. in a fasted state (water intake is permitted and encouraged). Upon arrival at the laboratory a trained phlebotomist staff member will insert a cannula (a small plastic tube) into a vein in the back of the hand. Participants will then be given one of the four test drinks, which once ingested will initiate the trial. Just after the ingestion of the test drink we will ask you to fill out a palatability scale.

Blood samples will be taken at baseline, and at 15, 30, 45, 60, 90, 120 and 180 minutes after ingestion of the test drink. An appetite questionnaire will also be completed at baseline and every 60 minutes after ingestion of the test drink to assess appetite sensations. After the 180-minute time point participants will be asked to consume a lunch meal until they are comfortably full. Once satisfied with the lunch meal they will fill out the final appetite questionnaire. The trial day will then be complete. Following study completion participants will be asked to complete a restrained eating questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 25.0-34.9 kg∙m-2
* Age 18-65 years
* Able and willing to provide informed consent and safely comply with study procedures
* Females to maintain record of regular menstrual cycle phase or contraceptive use
* No anticipated changes in diet/physical activity during the study (e.g. holidays or diet plans)

Exclusion Criteria:

* Allergies or adverse reactions to calcium or milk proteins.
* Contradictions to a high intake of calcium e.g. history of kidney stones
* Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias
* Any diagnosed metabolic disease (e.g. type 1 or type 2 diabetes)
* Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment
* Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)
* Any reported recent (<6 months) change in body mass (± 3%)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Total plasma glucagon-like peptide-1 concentrations | 4 hours
  Blood sampling

SECONDARY OUTCOMES:
Active plasma glucagon-like peptide-1 concentrations | 4 hours
  Blood sampling
Plasma insulin concentrations | 4 hours
  Blood sampling
Plasma NEFA concentrations | 4 hours
  Blood sampling
Plasma albumin concentrations | 4 hours
  Blood sampling
Serum calcium concentrations | 4 hours
  Blood sampling
Subjective appetite | 4 hours
  Visual appetite scales
ad libitum food intake | 4 hours
  lunch meal

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Health, University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Watkins JD, Smith HA, Hengist A, Brunsgaard LH, Mikkelsen UR, Koumanov F, Betts JA, Gonzalez JT. Plasma glucagon-like peptide-1 responses to ingestion of protein with increasing doses of milk minerals rich in calcium. Br J Nutr. 2021 Aug 9:1-9. doi: 10.1017/S000711452100297X. Online ahead of print. PMID 34369333